CLINICAL TRIAL: NCT07096427
Title: Effects of Health Promotion Model-Based Education Given to Pregnants With Virtual Reality on Healthy Living Behaviors
Brief Title: Virtual Reality-Based Health Promotion Education and Healthy Living Behaviors in Pregnant Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilgül Bacak, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024/36
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy; Health Behavior; Virtual Reality
Keywords: Pregnancy; Prenatal Education; Health Promotion; Health Promotion Behavior; Virtual Reality
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model in which participants are randomly assigned to one of three groups: (1) a virtual reality-based education group, (2) a booklet-based education group, or (3) a routine care control group. All interventions are delivered concurrently, and participants remain in their assigned group throughout the study period.
Who Masked: Participant
Masking Description: Participants were unaware of the group to which they were assigned (VR, booklet, or routine care). Researchers and outcome assessors were not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Education (Experimental): Participants receive education based on Pender's Health Promotion Model using virtual reality videos. The program includes three weekly sessions, each lasting about 20 minutes.
  Interventions: Behavioral: Virtual Reality-Based Prenatal Education
- Booklet-Based Education (Experimental): Participants receive the same educational content through printed booklets over three weekly face-to-face sessions of 20 minutes each.
  Interventions: Behavioral: Booklet-Based Prenatal Education
- Routine Care (No Intervention): Participants receive standard prenatal care provided at the Family Health Center. No additional educational intervention is applied.

INTERVENTIONS:
Behavioral: Virtual Reality-Based Prenatal Education — This intervention involves prenatal education based on Pender's Health Promotion Model delivered using immersive 360-degree virtual reality (VR) videos. The content focuses on healthy lifestyle behaviors during pregnancy, including nutrition, physical activity, stress management, and health responsibility. Participants view the videos via VR headsets in three weekly sessions, each lasting approximately 20 minutes. Motivational follow-up calls are conducted after the sessions.
  Arms: Virtual Reality Education
Behavioral: Booklet-Based Prenatal Education — This intervention includes prenatal education based on Pender's Health Promotion Model delivered through printed booklets. The educational content is identical to that of the VR group and covers healthy behaviors in pregnancy. The booklets are discussed in three face-to-face sessions, held once per week for three weeks. Each session lasts about 20 minutes. Participants receive motivational follow-up phone calls after the sessions.
  Arms: Booklet-Based Education

SUMMARY:
his study is a randomized controlled, single-blind, experimental research aiming to evaluate the effects of education based on Pender's Health Promotion Model-delivered through virtual reality (VR) technology and educational booklets-on healthy lifestyle behaviors in pregnant women. The study will be conducted in two Family Health Centers in Istanbul, and a total of 96 pregnant women will be randomly assigned to three groups: Experimental Group 1 (VR-based education), Experimental Group 2 (education with booklet), and Control Group (routine care). The experimental groups will receive three educational sessions, once a week for three weeks. Following the education sessions, motivational telephone interviews and follow-up assessments will be conducted. Data will be collected using the Healthy Lifestyle Behaviors in Pregnancy Scale (HLBPS), the Depression Anxiety Stress Scale (DASS-21), follow-up forms, and a postpartum evaluation form. The study aims to assess the effectiveness and sustainability of different educational methods on promoting healthy lifestyle behaviors among pregnant women.

DETAILED DESCRIPTION:
Pregnancy is a critical period that significantly alters a woman's lifestyle and necessitates the adoption of healthy behaviors. During pregnancy, engaging in healthy lifestyle behaviors such as attending regular prenatal checkups, avoiding harmful habits, maintaining a balanced diet, performing regular physical activity, and managing stress effectively is of great importance. Neglecting these behaviors can result in serious complications such as preterm birth, low birth weight, and the need for intensive care unit admission.

To support behavioral changes during this period, various behavior change theories are utilized. Among these, Pender's Health Promotion Model (HPM) evaluates cognitive, emotional, and environmental factors collectively to facilitate the development of health-promoting behaviors. The model explains the formation of health behaviors by considering individuals' previous experiences, perceived benefits and barriers, self-efficacy, and interpersonal influences.

The American College of Obstetricians and Gynecologists (ACOG) recommends the adequate intake of nutrients such as folic acid, iron, calcium, and vitamin D during pregnancy, along with increased water consumption and regular exercise. Exercise has been shown to reduce postpartum depression and accelerate recovery. Furthermore, ACOG emphasizes the importance of stress management and social support and recommends providing women with counseling services both during pregnancy and the postpartum period.

Nutrition education based on Pender's model has been shown to significantly improve diet quality in intervention groups. Similarly, interactive training materials such as role-play, simulations, and games have demonstrated a positive impact on pregnant women's health knowledge and behaviors.

This study will utilize two types of educational materials: virtual reality (VR) and printed educational booklets. VR provides individuals with a three-dimensional, interactive, and realistic learning environment, enhancing the effectiveness of health education. Studies have shown that VR reduces labor pain and anxiety and improves metabolic parameters in pregnant women with gestational diabetes.

There is a lack of comprehensive, theory-based, and technology-assisted interventions targeting behavioral change in pregnant women. Therefore, this study aims to evaluate the effectiveness of education delivered via VR and booklets-both based on Pender's model-on healthy lifestyle behaviors during pregnancy.

A total of 96 pregnant women will be randomly assigned to three groups:

Experimental Group 1: Three-session model-based education delivered via virtual reality headset.

Experimental Group 2: Three-session model-based face-to-face education using printed booklets.

Control Group: Routine prenatal care only. Data will be collected using the Healthy Lifestyle Behaviors in Pregnancy Scale (HLBPS), the Depression Anxiety Stress Scale (DASS-21), follow-up forms, and postpartum evaluation forms. After the intervention, motivational follow-up phone calls will be conducted. This study is expected to demonstrate the impact of a VR-based, evidence-informed educational program tailored to pregnant women on the adoption and sustainability of health-promoting behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 12-16 weeks of gestation
* Primigravida (first pregnancy)
* No chronic disease or health condition affecting lifestyle behaviors
* Able to communicate and give informed consent

Exclusion Criteria:

* High-risk pregnancies (e.g., gestational diabetes, preeclampsia, multiple pregnancy, threatened preterm labor)
* Existing psychiatric or communication impairments (e.g., language barrier)
* Having previously participated in similar educational programs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility to participate is based on biological sex (female), regardless of gender identity, due to the nature of the study targeting pregnant individuals.
Enrollment: 96 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Healthy Lifestyle Behaviors in Pregnancy | From baseline (12-16 weeks gestation) to follow-up (38 week gestation)
  The Healthy Lifestyle Behaviors in Pregnancy Scale is a 29-item, 5-point Likert-type instrument assessing six domains: pregnancy responsibility, hygiene, nutrition, physical activity, travel, and acceptance of pregnancy. Total scores range from 39 to 145, with higher scores reflecting healthier lifestyle behaviors during pregnancy.

SECONDARY OUTCOMES:
From baseline (12-16 weeks gestation) to follow-up (32-36 weeks gestation) | From baseline (12-16 weeks gestation) to follow-up (38 week gestation)
  The Depression Anxiety Stress Scale (DASS-21) is a 21-item self-report instrument that measures emotional states of depression, anxiety, and stress. It consists of three subscales with 7 items each. Items are rated on a 4-point Likert scale from 0 (never) to 3 (almost always). Higher scores indicate greater levels of emotional distress. The scale assesses symptoms experienced over the past week.

CONTACTS AND LOCATIONS:
Locations (1):
- Kagithane 13 Nolu Aile Sağlığı Merkezi, Istanbul, Kagithane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because data sharing was not included in the informed consent process.

REFERENCES:
- [Background] Estrella-Juarez F, Requena-Mullor M, Garcia-Gonzalez J, Lopez-Villen A, Alarcon-Rodriguez R. Effect of Virtual Reality and Music Therapy on the Physiologic Parameters of Pregnant Women and Fetuses and on Anxiety Levels: A Randomized Controlled Trial. J Midwifery Womens Health. 2023 Jan;68(1):35-43. doi: 10.1111/jmwh.13413. Epub 2022 Nov 16. PMID 36383473
- [Background] Jerald, J. (2015). The VR Book: Human-Centered Design for Virtual Reality. Morgan & Claypool.
- [Background] Permatasari TAE, Rizqiya F, Kusumaningati W, Suryaalamsah II, Hermiwahyoeni Z. The effect of nutrition and reproductive health education of pregnant women in Indonesia using quasi experimental study. BMC Pregnancy Childbirth. 2021 Mar 4;21(1):180. doi: 10.1186/s12884-021-03676-x. PMID 33663418
- [Background] Goodarzi-Khoigani M, Baghiani Moghadam MH, Nadjarzadeh A, Mardanian F, Fallahzadeh H, Mazloomy-Mahmoodabad S. Impact of Nutrition Education in Improving Dietary Pattern During Pregnancy Based on Pender's Health Promotion Model: A Randomized Clinical Trial. Iran J Nurs Midwifery Res. 2018 Jan-Feb;23(1):18-25. doi: 10.4103/ijnmr.IJNMR_198_16. PMID 29344041
- [Background] American College of Obstetricians and Gynecologists. (2023). Nutrition During Pregnancy. Retrieved from https://www.acog.org/womens-health/faqs/nutrition-during-pregnancy.
- [Background] Physical Activity and Exercise During Pregnancy and the Postpartum Period: ACOG Committee Opinion, Number 804. Obstet Gynecol. 2020 Apr;135(4):e178-e188. doi: 10.1097/AOG.0000000000003772. PMID 32217980
- [Background] Estebsari F, Dastoorpoor M, Mostafaei D, Khanjani N, Khalifehkandi ZR, Foroushani AR, Aghababaeian H, Taghdisi MH. Design and implementation of an empowerment model to prevent elder abuse: a randomized controlled trial. Clin Interv Aging. 2018 Apr 17;13:669-679. doi: 10.2147/CIA.S158097. eCollection 2018. PMID 29713151
- [Background] Mohamadian, H., Eftekhar Ardebili, H., Rahimi Foroushani, A., Taghdisi, M. H., & Shojaiezade, D. (2011). Evaluation of Pender's health promotion model for predicting adolescent girls' quality of life. Journal of School of Public Health & Institute of Public Health Research, 8(4).
- [Background] Malakouti J, Sehhati F, Mirghafourvand M, Nahangi R. Relationship between Health Promoting Lifestyle and Perceived Stress in Pregnant Women with Preeclampsia. J Caring Sci. 2015 Jun 1;4(2):155-63. doi: 10.15171/jcs.2015.016. eCollection 2015 Jun. PMID 26161369
- [Background] Lin YH, Tsai EM, Chan TF, Chou FH, Lin YL. Health promoting lifestyles and related factors in pregnant women. Chang Gung Med J. 2009 Nov-Dec;32(6):650-61. PMID 20035645